CLINICAL TRIAL: NCT01763333
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1026706 in Healthy Male Volunteers in a Partially Randomised, Single-blind, Placebo-controlled Trial, and Investigation of Relative Bioavailability of BI 1026706 (Open-label, Randomised, Four-way Cross-over)
Brief Title: To Investigate the Safety, Tolerability, Pharmacokinetics and the Relative Bioavailability of BI 1026706
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1320.1; 2012-002366-12 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-01-07; First posted 2013-01-08 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-12

CONDITIONS: Healthy

ARMS (2):
- 1 BI 1026706 single rising dose part (Experimental): single rising doses of BI 1026706
  Interventions: Drug: BI 1026706 Placebo; Drug: BI 1026706
- 2 BI 1026706 bioavailability part (Experimental): bioavailability part of BI 1026706
  Interventions: Drug: BI 1026706

INTERVENTIONS:
Drug: BI 1026706 Placebo — Placebo to BI 1026706
  Arms: 1 BI 1026706 single rising dose part
Drug: BI 1026706 — different dose formulations

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics and the relative bioavailability of BI 1026706

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2013-09-04 (Actual); Study Completion 2013-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1320.1.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the volunteers' pool of the Human Pharmacology Centre of Boehringer Ingelheim (BI) Pharma GmbH & Co. KG, Ingelheim, Germany.Only male subjects were included because no data on reproductive toxicology was available.
Pre-assignment Details: 68 subjects were randomised for single rising dose (SRD) part &12 subjects for bioavailability(BA) part of study.
Groups:
- BI 1026706 - Tablet 25 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 25 mg film coated tablet with 240 mL of water under fasted condition.
- BI 1026706 - Tablet 50 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 50 mg (2x25 mg) film coated tablet with 240 mL of water under fasted condition.
- BI 1026706 - Tablet 100 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 100 mg film coated tablet with 240 mL of water under fasted condition.
- BI 1026706 - Tablet 200 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 200 mg (2x100 mg) film coated tablet with 240 mL of water under fasted condition.
- BI 1026706 - Tablet 400 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 400 mg (4x100 mg) film coated tablet with 240 mL of water under fasted condition.
- BI 1026706 - Solution 10 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 10 mg solution under fasted condition.
- BI 1026706 - Solution 100 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 100 mg solution under fasted condition
- BI 1026706 - Solution 200 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 200 mg solution under fasted condition.
- BI 1026706 - Solution 400 mg (SRD - Part): Subjects were treated in the morning with one single oral dose of 400 mg solution under fasted condition.
- Placebo (SRD - Part): Subjects were treated in the morning with one single oral dose of matching placebo tablet and also matching placebo solution with 240 mL of water under fasted condition.
- R1/T1/R2/T2 (BA - Part): Subjects were treated in each of the 4 treatment periods with one single oral dose in the morning, First they were treated with 100mg film coated tablet (R1) under fasted condition, followed by 100mg film coated tablet (T1) under fed condition, 100 mg drinking solution (R2) under fasting and in the last treatment period with 100 mg drinking solution (T2) under fed condition. There was washout period of 7days between the respective treatments.
- T1/T2/R1/R2 (BA - Part): Subjects were treated in each of the 4 treatment periods with one single oral dose in the morning. First they were treated with 100mg film coated tablet (T1) under fed condition, followed by 100 mg drinking solution (T2) under fed condition, 100mg film coated tablet (R1) under fasted condition and in the last treatment period with 100 mg drinking solution (R2) under fasting condition. There was a washout period of 7days between the respective treatments.
- R2/R1/T2/T1 (BA - Part): Subjects were treated in each of the 4 treatment periods with one single oral dose in the morning, First they were treated with 100 mg drinking solution (R2) under fasting condition, followed by 100mg film coated tablet (R1) under fasted condition,100 mg drinking solution (T2) under fed condition and in the last treatment period with 100mg film coated tablet (T1) under fed condition. There was washout period of 7days between the respective treatments.
- T2/R2/T1/R1 (BA - Part): Subjects were treated in each of the 4 treatment periods with one single oral dose in the morning, First they were treated with 100 mg drinking solution (T2) under fed condition, followed by 100 mg drinking solution (R2) under fasting, 100mg film coated tablet (T1) under fed condition and in the last treatment period with 100mg film coated tablet (R1) under fasted condition. There was washout period of 7days between the respective treatments.
Period: Overall Study
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | Placebo (SRD - Part) | R1/T1/R2/T2 (BA - Part) | T1/T2/R1/R2 (BA - Part) | R2/R1/T2/T1 (BA - Part) | T2/R2/T1/R1 (BA - Part)
Started | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 18 | 3 | 3 | 3 | 3
Completed | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 18 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | Placebo (SRD - Part) | R1/T1/R2/T2 (BA - Part) | T1/T2/R1/R2 (BA - Part) | R2/R1/T2/T1 (BA - Part) | T2/R2/T1/R1 (BA - Part) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 18 | 3 | 3 | 3 | 3 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (4.2) | 39.0 (5.8) | 35.5 (7.1) | 39.5 (7.3) | 42.0 (5.7) | 39.7 (8.0) | 43.4 (7.8) | 35.7 (9.2) | 32.4 (12.0) | 35.9 (7.2) | 32.7 (12.4) | 27.0 (3.6) | 26.7 (4.9) | 27.0 (5.6) | 36.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 18 | 3 | 3 | 3 | 3 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug Related Adverse Events
Description: Percentage of subjects with drug related adverse events.
Time Frame: From the first dose of study medication upto 15 days after the day of last intake of study medication, upto 32 days for SRD Part and 30 days for BA Part.
Population: The treated set (TS) included all subjects who were documented to have taken at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Groups:
- BI 1026706 - Solution 100 mg Fasted (R2): Subjects were treated with 100 mg drinking solution (R2) under fasting condition.
- BI 1026706 - 100 mg Solution Fed (T2): Subjects were treated with 100 mg drinking solution (T2) under fed condition.
- BI 1026706 - Tablet 100 mg Fasted (R1): Subjects were treated with 100mg film coated tablet (R1) under fasted condition.
- BI 1026706 - Tablet 100 mg Fed (T1): Subjects were treated with 100mg film coated tablet (T1) under fed condition.
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | Placebo (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 18 | 11 | 12 | 12 | 10
Percentage of participants | 0.0 | 33.3 | 16.7 | 16.7 | 25.0 | 0.0 | 20.0 | 16.7 | 60.0 | 22.2 | 0.0 | 8.3 | 16.7 | 20.0

2. Secondary Outcome: Cmax
Description: Maximum measured concentration of the analyte in plasma (Cmax).
  The treated set-SRD Part (TS-SRD) included all 68 subjects from the TS who participated in the SRD Part. The treated set-BA Part (TS-BA) included all 12 subjects from the TS who participated in the BA Part.
  The per protocol set for the evaluation of relative bioavailability of T1 vs R1 (PPS-BA-T1-R1) included all subjects of the TS-BA who provided observations under the reference treatment (R1) or test treatment (T1) for at least one of the endpoints Cmax, AUC0-tz, or AUC0-inf,without experiencing emesis at or before two times median tmax and without important protocol violations (PVs) relevant to the statistical evaluation of pharmacokinetic (PK). The same definition applies for the analysis set PPS-BA-T2-R2, PPS-BA-R2-R1 and PPS-BA-T2-T1.
Time Frame: -2.0 hours (h) before dosing and 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: TS-SRD, TS-BA, PPS-DP, PPS-BA-T1-R1, PPS-BA-T2-R2, PPS-BA-R2-R1 and PPS-BA-T2-T1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles Per Litre (nmol/L)
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 11 | 12 | 12 | 10
nanomoles Per Litre (nmol/L) | 117 (33.1) | 268 (42.9) | 623 (40.9) | 728 (26.8) | 1430 (80.0) | 112 (32.9) | 1150 (47.1) | 2210 (28.0) | 3090 (24.8) | 1340 (32.0) | 706 (33.5) | 560 (34.8) | 651 (34.4)
Statistical Analysis 1: Comparison: BI 1026706 - Tablet 25 mg (SRD - Part) vs BI 1026706 - Tablet 50 mg (SRD - Part) vs BI 1026706 - Tablet 100 mg (SRD - Part) vs BI 1026706 - Tablet 200 mg (SRD - Part) vs BI 1026706 - Tablet 400 mg (SRD - Part); This was non confirmatory testing (Single dose). Dose proportionality of tablets for Cmax was analysed. The per protocol set for the evaluation of dose proportionality (PPS-DP) was used. This set included all subjects of the TS-SRD who provided at least one observation for at least one of the endpoints Cmax, AUC0-tz, AUC0-∞, or Aet1-t2, without experiencing emesis at or before 2 times median tmax and without important PVs relevant to the statistical evaluation of PK; Test type: Superiority or Other; Slope = 0.8728, 95% CI 2-sided [0.6942 to 1.0513] — Dose proportionality was explored using the power model (ANCOVA). The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale
Statistical Analysis 2: Comparison: BI 1026706 - Solution 10 mg (SRD - Part) vs BI 1026706 - Solution 100 mg (SRD - Part) vs BI 1026706 - Solution 200 mg (SRD - Part) vs BI 1026706 - Solution 400 mg (SRD - Part); This was non confirmatory testing (Single dose). Dose proportionality of solution for Cmax was analysed. The per protocol set for the evaluation of dose proportionality (PPS-DP) was used. This set included all subjects of the TS-SRD who provided at least one observation for at least one of the endpoints Cmax, AUC0-tz, AUC0-∞, or Aet1-t2, without experiencing emesis at or before 2 times median tmax and without important PVs relevant to the statistical evaluation of PK; Test type: Superiority or Other; Slope = 0.9341, 95% CI 2-sided [0.8277 to 1.0405] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BI 1026706 - Tablet 100 mg Fasted (R1) vs BI 1026706 - Tablet 100 mg Fed (T1); Relative bioavailability comparison Tab. fed (T1): Tab. fasted (R1) for Cmax. The per protocol set for the evaluation of relative bioavailability of T1 vs R1 (PPS-BA-T1-R1) was used; Test type: Non-Inferiority or Equivalence — The pharmacokinetic parameters were log transformed (natural logarithm) prior to fitting the ANOVA model. The difference between the expected means of the 2 treatments of interest for each pairwise comparison were estimated by the difference in the corresponding Least Square Means (point estimate) and two-sided 90% confidence intervals based on the t-distribution were computed. These quantities were then back-transformed to the original scale to give the point estimator (geometric mean); gMean ratio = 112.74, 90% CI 2-sided [95.579 to 132.993] — Adjusted gMean ratio
Statistical Analysis 4: Comparison: BI 1026706 - Solution 100 mg Fasted (R2) vs BI 1026706 - 100 mg Solution Fed (T2); Relative bioavailability comparison Sol. fed (T2) : Sol. fasted (R2) for Cmax. The per protocol set for the evaluation of relative bioavailability of T2 vs R2 (PPS-BA-T2-R2) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 52.66, 90% CI 2-sided [40.488 to 68.499] — Adjusted gMean ratio
Statistical Analysis 5: Comparison: BI 1026706 - Solution 100 mg Fasted (R2) vs BI 1026706 - Tablet 100 mg Fasted (R1); Relative bioavailability comparison Sol. fasted (R2): Tab. fasted (R1) for Cmax. The per protocol set for the evaluation of relative bioavailability of R2 vs R1 (PPS-BA-R2-R1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 239.63, 90% CI 2-sided [197.445 to 290.830] — Adjusted gMean ratio
Statistical Analysis 6: Comparison: BI 1026706 - 100 mg Solution Fed (T2) vs BI 1026706 - Tablet 100 mg Fed (T1); Relative bioavailability comparison Sol. fed (T2): Tab. fed (T1) for Cmax. The per protocol set for the evaluation of relative bioavailability of T2 vs T1 (PPS-BA-T2-T1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 105.47, 90% CI 2-sided [85.427 to 130.208] — Adjusted gMean ratio

3. Secondary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration)
Description: Time from dosing to maximum measured concentration (tmax).
Time Frame: -2.0h before dosing and 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: The treated set-SRD Part (TS-SRD) included all 68 subjects from the TS who participated in the SRD Part. The treated set-BA Part (TS-BA) included all 12 subjects from the TS who participated in the BA Part.
Measure: Median (Full Range); unit: hours
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 11 | 12 | 12 | 10
hours | 1.74 [0.75 to 4.07] | 1.51 [1.00 to 3.00] | 1.75 [0.73 to 4.02] | 1.25 [0.76 to 4.02] | 2.23 [1.00 to 3.00] | 0.63 [0.50 to 1.00] | 0.50 [0.50 to 0.76] | 0.75 [0.42 to 0.75] | 0.75 [0.42 to 1.00] | 0.52 [0.50 to 0.75] | 0.75 [0.50 to 1.00] | 1.74 [0.75 to 3.02] | 1.26 [0.50 to 2.00]

4. Secondary Outcome: AUC0-inf
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
Time Frame: -2.0h before dosing and 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: TS-SRD, TS-BA, PPS-DP, PPS-BA-T1-R1, PPS-BA-T2-R2, PPS-BA-R2-R1 and PPS-BA-T2-T1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 11 | 12 | 12 | 10
nmol*h/L | 768 (28.6) | 1690 (51.8) | 3990 (30.9) | 4040 (29.4) | 8900 (85.1) | 428 (41.9) | 3220 (43.5) | 7790 (26.9) | 11300 (28.3) | 4590 (33.1) | 3380 (28.6) | 3270 (28.3) | 2930 (40.8)
Statistical Analysis 1: Comparison: BI 1026706 - Tablet 25 mg (SRD - Part) vs BI 1026706 - Tablet 50 mg (SRD - Part) vs BI 1026706 - Tablet 100 mg (SRD - Part) vs BI 1026706 - Tablet 200 mg (SRD - Part) vs BI 1026706 - Tablet 400 mg (SRD - Part); This was non confirmatory testing (Single dose).Dose proportionality of tablets for AUC0-inf was analysed.The per protocol set for the evaluation of dose proportionality (PPS-DP) was used. This set included all subjects of the TS-SRD who provided at least one observation for at least one of the endpoints Cmax, AUC0-tz, AUC0-∞, or Aet1-t2, without experiencing emesis at or before 2 times median tmax and without important PVs relevant to the statistical evaluation of PK; Test type: Superiority or Other; Slope = 0.8341, 95% CI 2-sided [0.6485 to 1.0198] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 1026706 - Solution 10 mg (SRD - Part) vs BI 1026706 - Solution 100 mg (SRD - Part) vs BI 1026706 - Solution 200 mg (SRD - Part) vs BI 1026706 - Solution 400 mg (SRD - Part); This was non confirmatory testing (Single dose).Dose proportionality of solution for AUC0-inf was analysed. The per protocol set for the evaluation of dose proportionality (PPS-DP) was used. This set included all subjects of the TS-SRD who provided at least one observation for at least one of the endpoints Cmax, AUC0-tz, AUC0-∞, or Aet1-t2, without experiencing emesis at or before 2 times median tmax and without important PVs relevant to the statistical evaluation of PK; Test type: Superiority or Other; Slope = 0.9149, 95% CI 2-sided [0.8059 to 1.0239] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BI 1026706 - Tablet 100 mg Fasted (R1) vs BI 1026706 - Tablet 100 mg Fed (T1); Relative bioavailability comparison Tab. fed (T1): Tab. fasted (R1) for AUC0-inf. The per protocol set for the evaluation of relative bioavailability of T1 vs R1 (PPS-BA-T1-R1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean Ratio = 86.61, 90% CI 2-sided [76.529 to 98.029] — Adjusted gMean ratio
Statistical Analysis 4: Comparison: BI 1026706 - Solution 100 mg Fasted (R2) vs BI 1026706 - 100 mg Solution Fed (T2); Relative bioavailability comparison Sol. fed (T2) : Sol. fasted (R2) for AUC0-inf.The per protocol set for the evaluation of relative bioavailability of T2 vs R2 (PPS-BA-T2-R2) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 74.44, 90% CI 2-sided [66.322 to 83.562] — Adjusted gMean ratio
Statistical Analysis 5: Comparison: BI 1026706 - Solution 100 mg Fasted (R2) vs BI 1026706 - Tablet 100 mg Fasted (R1); Relative bioavailability comparison Sol. fasted (R2): Tab. fasted (R1) for AUC0-inf.The per protocol set for the evaluation of relative bioavailability of R2 vs R1 (PPS-BA-R2-R1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 137.25, 90% CI 2-sided [119.708 to 157.353] — Adjusted gMean ratio
Statistical Analysis 6: Comparison: BI 1026706 - 100 mg Solution Fed (T2) vs BI 1026706 - Tablet 100 mg Fed (T1); Relative bioavailability comparison Sol. fed (T2): Tab. fed (T1) for AUC0-inf.The per protocol set for the evaluation of relative bioavailability of T2 vs T1 (PPS-BA-T2-T1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 116.48, 90% CI 2-sided [111.462 to 121.724] — Adjusted gMean ratio

5. Secondary Outcome: AUC0- tz
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0- tz).
Time Frame: -2.0h before dosing and 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: TS-SRD, TS-BA, PPS-DP, PPS-BA-T1-R1, PPS-BA-T2-R2, PPS-BA-R2-R1 and PPS-BA-T2-T1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 11 | 12 | 12 | 10
nmol*h/L | 741 (25.2) | 1670 (51.8) | 3950 (30.5) | 3990 (28.6) | 8830 (85.3) | 403 (44.0) | 3170 (27.0) | 7710 (27.0) | 11300 (28.3) | 4550 (33.3) | 3360 (28.9) | 3240 (28.3) | 2900 (40.8)
Statistical Analysis 1: Comparison: BI 1026706 - Tablet 25 mg (SRD - Part) vs BI 1026706 - Tablet 50 mg (SRD - Part) vs BI 1026706 - Tablet 100 mg (SRD - Part) vs BI 1026706 - Tablet 400 mg (SRD - Part); This was non confirmatory testing (Single dose). Dose proportionality of tablets for AUC 0- tz was analysed. The per protocol set for the evaluation of dose proportionality (PPS-DP) was used. This set included all subjects of the TS-SRD who provided at least one observation for at least one of the endpoints Cmax, AUC0-tz, AUC0-∞, or Aet1-t2, without experiencing emesis at or before 2 times median tmax and without important PVs relevant to the statistical evaluation of PK; Test type: Superiority or Other; Slope = 0.8428, 95% CI 2-sided [0.6580 to 1.0275] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: BI 1026706 - Solution 10 mg (SRD - Part) vs BI 1026706 - Solution 100 mg (SRD - Part) vs BI 1026706 - Solution 200 mg (SRD - Part) vs BI 1026706 - Solution 400 mg (SRD - Part); This was non confirmatory testing (Single dose). Dose proportionality of solution for AUC0-tz was analysed. The per protocol set for the evaluation of dose proportionality (PPS-DP) was used. This set included all subjects of the TS-SRD who provided at least one observation for at least one of the endpoints Cmax, AUC0-tz, AUC0-∞, or Aet1-t2, without experiencing emesis at or before 2 times median tmax and without important PVs relevant to the statistical evaluation of PK; Test type: Superiority or Other; Slope = 0.9307, 95% CI 2-sided [0.8187 to 1.0426] — Dose proportionality was explored using the power model (ANCOVA). The perfect dose proportionality would correspond to a slope β of 1
Statistical Analysis 3: Comparison: BI 1026706 - Tablet 100 mg Fasted (R1) vs BI 1026706 - Tablet 100 mg Fed (T1); Relative bioavailability comparison Tab. fed (T1) : Tab. fasted (R1) for AUC 0-tz. The per protocol set for the evaluation of relative bioavailability of T1 vs R1 (PPS-BA-T1-R1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean Ratio = 86.16, 90% CI 2-sided [75.735 to 98.027] — Adjusted geometric mean (gMean) ratio
Statistical Analysis 4: Comparison: BI 1026706 - Solution 100 mg Fasted (R2) vs BI 1026706 - 100 mg Solution Fed (T2); Relative bioavailability comparison Sol. fed (T2) : Sol. fasted (R2) for AUC 0-tz.The per protocol set for the evaluation of relative bioavailability of T2 vs R2 (PPS-BA-T2-R2) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 74.42, 90% CI 2-sided [65.979 to 83.941] — Adjusted gMean ratio
Statistical Analysis 5: Comparison: BI 1026706 - Solution 100 mg Fasted (R2) vs BI 1026706 - Tablet 100 mg Fasted (R1); Relative bioavailability comparison Sol. fasted (R2): Tab. fasted (R1) for AUC 0-tz.The per protocol set for the evaluation of relative bioavailability of R2 vs R1(PPS-BA-R2-R1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 137.20, 90% CI 2-sided [119.611 to 157.374] — Adjusted gMean ratio
Statistical Analysis 6: Comparison: BI 1026706 - 100 mg Solution Fed (T2) vs BI 1026706 - Tablet 100 mg Fed (T1); Relative bioavailability comparison Sol. fed (T2): Tab. fed (T1) for AUC 0-tz.The per protocol set for the evaluation of relative bioavailability of T2 vs T1 (PPS-BA-T2-T1) was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; gMean ratio = 116.83, 90% CI 2-sided [111.814 to 122.079] — Adjusted gMean ratio

6. Secondary Outcome: t1/2 (Terminal Half-life of the Analyte in Plasma)
Description: Terminal half-life of the analyte in plasma (t1/2).
Time Frame: -2.0h before dosing and 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after dosing
Population: TS-SRD and TS-BA
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 5 | 11 | 12 | 12 | 10
hours | 10.80 (75.7) | 8.58 (54.3) | 12.10 (26.6) | 11.60 (43.2) | 12.00 (22.7) | 13.90 (82.1) | 12.80 (54.7) | 11.50 (50.3) | 9.29 (27.3) | 10.80 (36.0) | 11.10 (53.9) | 10.50 (46.9) | 12.60 (28.4)

7. Secondary Outcome: f t1-t2 (SRD-Part)
Description: Fraction of analyte eliminated in urine from the time point t1 (0h) to time point t2 (72h) (f t1-t2).
Time Frame: 0-4, 4-8, 8-12, 12-24, 24-48, 48-72 hours
Population: TS-SRD
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 4 | 6 | 5 | 6 | 5
Percentage | 3.02 (21.1) | 2.75 (51.2) | 3.43 (33.4) | 1.95 (27.2) | 1.87 (45.3) | 3.97 (40.8) | 3.47 (23.9) | 3.82 (32.8) | 2.09 (7.44)

ADVERSE EVENTS:
Time Frame: From the first dose of study medication upto 15 days after the day of last intake of study medication, upto 32 days for SRD Part and 30 days for BA Part.
Arm/Group | BI 1026706 - Tablet 25 mg (SRD - Part) | BI 1026706 - Tablet 50 mg (SRD - Part) | BI 1026706 - Tablet 100 mg (SRD - Part) | BI 1026706 - Tablet 200 mg (SRD - Part) | BI 1026706 - Tablet 400 mg (SRD - Part) | BI 1026706 - Solution 10 mg (SRD - Part) | BI 1026706 - Solution 100 mg (SRD - Part) | BI 1026706 - Solution 200 mg (SRD - Part) | BI 1026706 - Solution 400 mg (SRD - Part) | Placebo (SRD - Part) | BI 1026706 - Solution 100 mg Fasted (R2) | BI 1026706 - 100 mg Solution Fed (T2) | BI 1026706 - Tablet 100 mg Fasted (R1) | BI 1026706 - Tablet 100 mg Fed (T1)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/5 | 0/6 | 0/5 | 0/18 | 0/11 | 0/12 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 5/6 | 3/6 | 2/6 | 2/4 | 3/6 | 2/5 | 1/6 | 4/5 | 8/18 | 3/11 | 3/12 | 6/12 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1026706 - Tablet 25 mg (SRD - Part) (N=6) | BI 1026706 - Tablet 50 mg (SRD - Part) (N=6) | BI 1026706 - Tablet 100 mg (SRD - Part) (N=6) | BI 1026706 - Tablet 200 mg (SRD - Part) (N=6) | BI 1026706 - Tablet 400 mg (SRD - Part) (N=4) | BI 1026706 - Solution 10 mg (SRD - Part) (N=6) | BI 1026706 - Solution 100 mg (SRD - Part) (N=5) | BI 1026706 - Solution 200 mg (SRD - Part) (N=6) | BI 1026706 - Solution 400 mg (SRD - Part) (N=5) | Placebo (SRD - Part) (N=18) | BI 1026706 - Solution 100 mg Fasted (R2) (N=11) | BI 1026706 - 100 mg Solution Fed (T2) (N=12) | BI 1026706 - Tablet 100 mg Fasted (R1) (N=12) | BI 1026706 - Tablet 100 mg Fed (T1) (N=10)
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 3 | 1 | 1 | 3 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes